CLINICAL TRIAL: NCT05620810
Title: Neuropsychiatric Symptoms in Spontaneous Intracerebral Hemorrhage Survivors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202210006RIND
Record Dates: First submitted 2022-11-11; First posted 2022-11-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-10

CONDITIONS: Primary Disease or Condition Being Studied, or Focus of the Study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: neuropsychiatric symptoms — neuropsychiatric symptoms

SUMMARY:
Compared to the United Kingdom and the United States, Spontaneous non-traumatic intracerebral hemorrhage (ICH) is more common among people in Taiwan. The prevalence rate of ICH was 14.0% for people aged 36 years or older in Taiwan. Primary ICH originates from the spontaneous rupture of small vessels damaged by chronic hypertension or cerebral amyloid angiopathy (CAA). Emotional disturbances are frequent symptoms in stroke survivors and negatively impact on functional recovery, the patient's quality of life and are distressing for both the patients and their caregivers. Furthermore, the emotional disturbances are associated with impaired cognitive. However, these issues are often unnoticed and most of the studies had been performed in ischemic stroke survivors rather than in patients with ICH.

In this study, we will be recruited participants from National Taiwan University Hospital Bei-Hu branch and National Taiwan University Hospital. We aim to enroll respectively maximum number of 60 patients who had previous spontaneous ICH. Each participant will receive neuropsychiatric assessment, cognitive screening tests, domain-specific cognitive tests, a questionnaire for their quality of life and blood drawing for ApoE genotyping. The main aims of this study include (1) To investigate the prevalence of distinct neuropsychiatric symptoms in ICH survivors (2) To investigate the impact of non-cognitive neuropsychiatric issues on the cognitive functions and quality of life in ICH survivors. Our results may remind clinicians to pay more attention to the early diagnosis and effective management of neuropsychiatric symptoms to improve clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is older than 20-year-old (older than 18-year-old from Jan 1st, 2023) with a past medical history of spontaneous intracerebral hemorrhage.
2. The weight of patient is over 50 Kilograms
3. Patient agrees to participate in the study

Exclusion Criteria:

1. Patients who experience acute phase of stroke or neurological disorders, or vision loss and hearing impairment
2. Patient cannot cooperate with the interview including those with aphasia, conscious disturbance or bedridden status

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be recruited participants from National Taiwan University Hospital Bei-Hu branch and National Taiwan University Hospital Neurology Clinic. We aim to enroll respectively maximum number of 60 patients who had previous spontaneous ICH.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
To investigate the prevalence of distinct neuropsychiatric symptoms in ICH survivors | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Bei-Hu Branch, National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided